CLINICAL TRIAL: NCT01149031
Title: Low Level Laser Therapy for the Treatment of Provoked Vestibulodynia
Acronym: LLLT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, Clinic for vulvovaginal disorders, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ahinoam110-HMO-CTIL
Record Dates: First submitted 2010-06-16; First posted 2010-06-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Provoked Vestibulodynia
Keywords: Provoked Vestibulodynia; Low Level Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- low level laser therapy, using a probe (Active Comparator): The treatment will be done by using a LLL-probe touching several areas of the vulvar vestibule, according to the selected protocol.
  Every patient will be treated twice weekly for 6 weeks.
  Interventions: Device: LOW LEVEL LASER SYSTEM
- Placebo (Placebo Comparator): The patients will be treated with placebo-probe, according to the same protocol
  Interventions: Device: LOW LEVEL LASER SYSTEM

INTERVENTIONS:
Device: LOW LEVEL LASER SYSTEM — LASER DIODE CLASS 3B,OMEGA XP
  Other Names: LASER DIODE CLASS 3B,OMEGA XP

SUMMARY:
Provoked vestibulodynia, previously called vulvar vestibulitis syndrome, is clinically defined as chronic, unexplained, vulvar pain or discomfort confined to the vulvar vestibule in response to contact or pressure. In addition, many patients also have pain in response to non-sexual activities such as tampon insertion, gynecological examinations or physical pursuits such as bicycle riding; the severity of other vulvo-vaginal symptoms such as itching, burning and irritation varies. Once women with provoked vestibulodynia develop the syndrome, symptoms may last for months or years; as a result, provoked vestibulodynia has a profound effect on women's sexuality and psychological well-being. The diagnosis of provoked vestibulodynia is usually made by ascertaining if the patient fulfills modified Friedrich's criteria, consisting of 1) a history of vulvar pain, dyspareunia or pain with tampon insertion, 2) tenderness of the vestibule when being touched with a cotton-tip applicator and 3) no identifiable cause for the pain.

The etiology of this condition remains unknown. Proposed causes include chronic inflammation, peripheral neuropathy, genetic, immunologic and hormonal factors, infectious, psychological disorders, sexual dysfunction or disturbance in the central nervous system. Because the cause of provoked vestibulodynia remains unknown, many different treatments have been described for this condition, including topical and intra-lesional corticosteroids, topical anesthetics such as lidocaine, topical estrogen, topical or oral antidepressants or anti-convulsants, biofeedback or physical therapy, surgical resection of the involved tissue (vestibulectomy) and a variety of complementary and alternative therapies.

Low level laser therapy (LLLT) is an emerging medical technique in which exposure to low-level laser light or light emitting diodes might stimulate or inhibit cellular function, possibly leading to beneficial clinical effects. Clinical applications that show some potential of effectiveness include treating soft tissue injury, chronic pain, and wound healing. The usage of low level laser therapy was found effective in various pain syndromes, and has no side effects.

Since inflammatory mechanisms have been proposed in the pathogenesis of provoked vestibulodynia, and as there is no effective therapy for this syndrome, the investigators intend to study whether low level laser therapy might be an effective therapy for provoked vestibulodynia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with provoked vestibulodynia who meet modified Friedrich's criteria, after exclusion of other vulvar disorders, who are willing to participate in the study.

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in vestibular pain level(as measured by variable parameters) | 7 weeks (at the end of treatment protocol)
  Response to treatment will be assessed by change in pain by numeric rating scale of a weekly Tampon Test, change in overall daily pain intensity (24 hour numeric rating scale), frequency of sexual intercourse, the change in intercourse pain numeric rating scale, and the cotton swab test pain level by verbal reporting scale. In addition, patients will complete quality-of-life questionnaires (Brief Pain Inventory and Neuropathic Pain Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev-Sagie, MD, Principal Investigator — Hadassah Medical Organization, Jerusalem
Locations (1):
- Ahinoam Lev-Sagie, Jerusalem, Israel